CLINICAL TRIAL: NCT05094674
Title: Clinical Validation of Biosafety Technologies Breath Analyser Tests for the Diagnosis of COVID-19; the Project Aims to Validate the Diagnostic Device and to Assess the Comparative Performance With RT-PCR Currently Being Deployed in the NHS.
Brief Title: Clinical Validation of Breath Analyser Tests for Diagnosis of COVID-19.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tera Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BREATHE
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The participant's breath sample is taken by blowing preferably three times into a disposable TeraTube. Thereafter, the tube is sealed, sterilized, and scanned by the BioSafety Station for analysis of its bio-chemical spectral signature. This will take place once during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants who require a diagnostic or screening COVID-19 RT-PCR test (Other): Participants who require a diagnostic or screening COVID-19 RT-PCR test, presenting at Tameside and Glossop Integrated Care NHS Foundation Trust aged 18 years or over
  Interventions: Diagnostic Test: Breath Sample analysis

INTERVENTIONS:
Diagnostic Test: Breath Sample analysis — The participant's breath sample is taken by blowing preferably three times into a disposable tube. Thereafter, the tube is sealed, sterilized, and scanned by the BioSafety Station for analysis. This will take place once during the study.

SUMMARY:
The Sponsor has developed a rapid screening tool intended to determine if the subject tested is COVID-19-free (Negative to COVID-19).

DETAILED DESCRIPTION:
Within this proposed project, the NHS will collect two diagnostic or screening tests per participant. One sample will be used by NHS and be run through regular diagnostics. The second, will be breath sample which will be tested using the BioSafety Technologies Ltd, rapid screening tool. This will use a pre-defined protocol. These tests would then be compared to assess the diagnostic efficacy including sensitivity and specificities. We will be aiming to achieve a significant comparison to ensure certainty and to exploit the information for proposing a novel diagnostic system to enhance capabilities to scale up the testing of patients. The proposed activity involves clinical validation of BioSafety Testing, to enhance the performance of detection along with clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Requiring a diagnostic or screening RT-PCR test for COVID-19

Exclusion Criteria:

* Subjects under general anaesthesia
* The inability to personally sign the consent form.
* The inability to exhale breath

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-06-22 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of positive and negative cases in collected breath samples using breath analyser test. | The collection of an additional samples requiring COVID 19 diagnostic evaluation will take approximately 1 minute from initial collection of the sample

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Lieberman, MD, Principal Investigator — Tameside and Glossop Integrated Care NHS England
Locations (1):
- Tameside and Glossop Integrated Care NHS, Ashton-under-Lyne, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No